CLINICAL TRIAL: NCT00470626
Title: Prospective Study of the Cook Celect Filter, Including Permanent and Retrievable Use
Brief Title: Celect Vena Cava Filter Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cook Group Incorporated (Industry)
Collaborators: MED Institute, Incorporated (Industry); William Cook Australia (Industry); William Cook Europe (Industry); Cook Ireland, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05-507; 110006, GTMX
Record Dates: First submitted 2005-09-14; First posted 2007-05-08 (Estimated); Results first posted 2010-04-06 (Estimated); Last update posted 2016-01-25 (Estimated); Status verified 2015-12

CONDITIONS: Pulmonary Embolism; Venous Thromboembolism
Keywords: Pulmonary Embolism; Venous Thromboembolism; Inferior Vena Cava Filter; IVC; PE
MeSH Terms: conditions — Pulmonary Embolism; Venous Thromboembolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Vena Cava Filter
  Interventions: Device: Celect Vena Cava Filter

INTERVENTIONS:
Device: Celect Vena Cava Filter — Effective filtration of inferior vena cava blood to prevent thromboembolism.

SUMMARY:
The clinical study will collect data to verify the safety and performance of the Cook Celect Filter in the prevention of pulmonary embolism (PE) in patients with a temporary or permanent high risk of thromboembolism.

ELIGIBILITY:
Inclusion Criteria:

* The patient is at high risk for pulmonary embolism and is under consideration for placement of a permanent or short-term IVC filter.
* The patient must have a patent internal jugular vein.
* The patient or guardian must have given informed consent.
* The patient must agree to return for clinical imaging follow-up at 1, 3, 6, and 12 months.
* The patient must agree to have a clinical and imaging examination performed prior to filter retrieval.
* The patient must agree to return for clinical and imaging follow-up at 30 days and 3 months after filter retrieval.

Exclusion Criteria:

* The patient is less than 18 years of age.
* The patient is pregnant.
* The patient has uncontrollable coagulopathy.
* The patient has a life expectancy less than 6 months.
* The patient has a vena cava diameter over 30 mm, measured by vena cava sizing catheters.
* The patient's vena cava diameter is less than 15 mm, measured by vena cava sizing catheters.
* The patient has a contrast allergy that can not be adequately pre-medicated.
* The patient is simultaneously participating in another investigative drug or device study, or has a previous IVC filter.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2005-11; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: R.W. Gunther, Prof., Principal Investigator — Klinik Fur Radiologische Diagnostik Universitaetklinikum der RWTH Aachen
Locations (8):
- The Alfred Hospital, Melbourne, Australia
- RWTH Aachen University, Aachen, Germany
- Mexico (2):
  - Instituto Nacional de Enfermedades Respiratorias, Mexico City
  - Hospital Universitario de Nuevo Leon, Monterrey
- Universitario Zaragoza - Hospital Clinico, Zaragoza, Spain
- United Kingdom (3):
  - North Hampshire Hospital, Hampshire
  - Leeds Teaching Hospitals NHS Trust, Leeds
  - John Radcliffe Hospital, Oxford

REFERENCES:
- [Result] Lyon SM, Riojas GE, Uberoi R, Patel J, Lipp ME, Plant GR, De Gregorio MA, Gunther RW, Voorhees WD, McCann-Brown JA. Short- and long-term retrievability of the Celect vena cava filter: results from a multi-institutional registry. J Vasc Interv Radiol. 2009 Nov;20(11):1441-8. doi: 10.1016/j.jvir.2009.07.038. PMID 19875061

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Celect Vena Cava Filter
Started | 129
Completed | 112
Not Completed | 17
Not completed — Lost to Follow-up | 10
Not completed — Withdrawal by Subject | 7

BASELINE CHARACTERISTICS:
Arm/Group | Celect Vena Cava Filter
Number analyzed (Participants) | 129
Age, Continuous [Mean (Standard Deviation); unit: years] | 51 (19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58
  Male | 71
Cancer [Number; unit: participants]
  Cancer | 23
  No Cancer | 106
Coagulation Disorder [Number; unit: participants]
  Coagulation Disorder | 4
  No Coagulation Disorder | 125
Congestive Heart Failure (CHF) [Number; unit: participants]
  CHF | 1
  No CHF | 128
Coronary Heart Disease (CHD) [Number; unit: participants]
  CHD | 1
  No CHD | 128
Current Deep Venous Thrombosis (DVT) [Number; unit: participants]
  Current DVT | 72
  No Current DVT | 57
Current Pulmonary Embolism (PE) [Number; unit: participants]
  Current PE | 50
  No Current PE | 79
Diabetes [Number; unit: participants]
  Diabetes Type I | 2
  Diabetes Type II | 10
  No Diabetes | 117
Gastrointestinal (GI) Disease [Number; unit: participants]
  GI Disease | 8
  No GI Disease | 121
Hepatic Disease [Number; unit: participants]
  Hepatic Disease | 3
  No Hepatic Disease | 126
Hypertension [Number; unit: participants]
  Hypertension | 0
  No Hypertension | 129
Peripheral Vascular Disease (PVD) [Number; unit: participants]
  PVD | 7
  No PVD | 122
Pulmonary Disease [Number; unit: participants]
  Pulmonary Disease | 33
  No Pulmonary Disease | 96
Renal Disease [Number; unit: participants]
  Renal Disease | 5
  No Renal Disease | 124
Stroke [Number; unit: participants]
  Stroke | 7
  No Stroke | 122
Trauma [Number; unit: participants]
  Trauma | 38
  No Trauma | 91

OUTCOME MEASURES:

1. Primary Outcome: Major Adverse Event
Description: Composite Major Adverse Event includes hemorrhage, perforation, pulmonary embolism, procedure-related or device-related death, occlusion, significant migration and filter fracture.
Time Frame: up to 12 months
Measure: Number; unit: participants
Arm/Group | Celect Vena Cava Filter
Number analyzed (Participants) | 129
participants
  Hemorrhage, Perforation | 0
  Pulmonary Embolism | 1
  Procedure or Device-Related Death | 2
  Inferior Vena Cava Occlusion | 0
  Significant Migration | 0
  Filter Fracture | 0

2. Secondary Outcome: Successful Retrieval
Description: Retrieval attempt describes a procedure in which a physician tried to remove a filter from a patient. A decision to remove a filter was made after determining that the patient no longer required the filter. Retrieval attempts were either successful (i.e., the filter was removed) or unsuccessful (i.e., the filter could not be removed and remained in the patient as a permanent device).
Time Frame: up to 12 months
Population: 129 patients received a filter. Filters were placed as permanent devices in 34 patients and as temporary devices in 95 patients. A decision to retrieve a filter was made by the physician once the patient's medical condition warranted it (once the fliter was no longer required). Filter retrieval was attempted in 58 of 95 patients.
Measure: Number; unit: successful retrievals
Arm/Group | Celect Vena Cava Filter
Number analyzed (Participants) | 58
successful retrievals | 56
Statistical Analysis 1: Comparison: Celect Vena Cava Filter; Test type: Superiority or Other; Probability of Successful Retrieval = .9 — Probability of successful retrieval is from Kaplan-Meier analysis

3. Secondary Outcome: Mean Time to Retrieval Attempt
Description: Mean time to retrieval describes the average time filters were in place in the study group before a retrieval attempt was made.
  A retrieval attempt describes a procedure in which a physician tried to remove a filter from a patient. The mean time to retrieval describes the average time filters were in place before a retrieval attempt was made.
Time Frame: up to 12 months
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Celect Vena Cava Filter
Number analyzed (Participants) | 58
days | 186 (124)

ADVERSE EVENTS:
Arm/Group | Celect Vena Cava Filter
Serious Adverse Events (participants affected / at risk) | 3/129
Other Adverse Events (participants affected / at risk) | 0/129
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Celect Vena Cava Filter (N=129)
Hemorrhage, Perforation (Injury, poisoning and procedural complications) | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1
Procedure or Device Related Death (Injury, poisoning and procedural complications) | 2 — 1 death occured within 24 hours of device placement. Poor overall health likely contributed to death. 1 death occurred 185 days post-procedure and was the result of a pulmonary thromboembolism; the location of the origin of the clot was unknown.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days